CLINICAL TRIAL: NCT03742544
Title: Post Marketing Surveillance of Telostop TAB (Telmisartan/Rosuvastatin) for Evaluating the Safety and Efficacy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ID-TERO-401
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Hypertension; Dyslipidemias
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Post-marketing surveillance of Telostop TAB (Telmisartan/Rosuvastatin)

DETAILED DESCRIPTION:
Telostop TAB is fixed-dose combination of telmisartan and rosuvastatin, which was approved in 2015 in the Republic of Korea for the treatment of patients with hypertention and dyslipidemia. A post-marketing surveillance was conducted following the approval to obtain data on the safety and efficacy of Telostop TAB in real-world practice.

ELIGIBILITY:
Inclusion Criteria:

* The patient who is first prescribed and administered Telostop plus Tab.

Exclusion Criteria:

* The patients who are overreacting to this drug or its components
* The patients to the "Do not administer to the next patient" section of the approved instructions for use

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: residents of Korea, in real-world practice
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-06-23 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse event after this drug administration in general medical practice | 24 weeks
  Any adverse events occurred after this drug dosing will be recorded. Description of adverse event(s) including type of adverse event(s), onset/end date, severity, action taken, causal relationship to the drug and investigator's view on the adverse event(s) will be captured, whether it is related to the drug or not and until follow up visit more than 1 time during the surveillance period.
  Lab abnormalities and changes in vital signs are considered to be adverse events only if they result in discontinuation from the study, necessitate therapeutic medical intervention, and/or if the investigator considers them to be adverse events.

SECONDARY OUTCOMES:
The change from baseline to week 24 in the LDL cholesterol | 24 weeks
  LDL cholesterol is measured before administration of the drug and within 24 weeks after administration.
The change from baseline to week 24 in the blood pressure | 24 weeks
  Blood pressure is measured before administration of the drug and within 24 weeks after administration.

IPD SHARING:
Plan to Share IPD: Undecided